CLINICAL TRIAL: NCT00256347
Title: Development of Analgesic Tolerance to Repeated Doses of Subcutaneous Morphine Using the Brief Thermal Sensitization Model in Healthy Volunteers
Brief Title: Analgesic Tolerance to Repeated Doses of Subcutaneous Morphine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: H5612-25135; H5612-25135
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-03

CONDITIONS: Healthy Volunteers

INTERVENTIONS:
Drug: intramuscular injections of morphine

SUMMARY:
30 healthy volunteers will be enrolled in this 6-session study. The first visit will be a screening/orientation session. The next 5 visits will be (full day) outpatient sessions taking place Monday through Friday during one week. All full day visits will be drug administration sessions with subjects randomized to one of two groups. The primary purpose is to investigate the time course of development of analgesic tolerance (loss of pain relieving effect) to morphine on experimentally produced skin tenderness in healthy volunteers.

DETAILED DESCRIPTION:
30 healthy volunteers will be enrolled in this 6-session study. The first visit will be a screening/orientation session. The next 5 visits will be (full day) outpatient sessions taking place Monday through Friday during one week. All full day visits will be drug administration sessions with subjects randomized to one of two groups. Group A will receive two daily intramuscular injections of 8 mg morphine on Monday through Thursday and two intramuscular injections of placebo on Friday. Group B will receive two daily intramuscular injections of placebo on Monday through Thursday and two intramuscular injections of 8 mg morphine on Friday. During the Monday through Friday sessions the painfulness of experimental heat application and the area of skin tenderness (primary and secondary hyperalgesia) will be assessed before and two times after the intramuscular injections. Heat will be applied by using a computer controlled probe that applies heat (450 C/1130 F) on the thigh for 3 minutes (Brief Thermal Sensitization model.)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers who are 21-50 years of age,
2. If female, must be non-lactating, not pregnant, and using a reliable contraception method (i.e. abstinence, intrauterine device [IUD], hormonal birth control, or double barrier method [male condom, female condom, or diaphragm plus a spermicidal agent such as contraceptive foam, jelly or cream]).
3. In stable health
4. Must weigh between 110 and 200 lbs and have a Body Mass Index between 20 and 30.
5. Able and willing to provide written informed consent
6. Able to understand and follow the instructions of the investigator, including the pain intensity rating scales
7. Develops temporary secondary hyperalgesia from the brief thermal sensitization stimulation procedure performed at the screening visit (Session 1)
8. Opioid naïve (no previous history of long term opioid use)

Exclusion Criteria:

1. Severe coronary artery disease, uncontrolled hypertension, cardiac ventricular conduction abnormalities, or orthostatic mean blood pressure drop > than 25 mmHg, severe chronic obstructive pulmonary disease.
2. History of renal or hepatic failure.
3. Evidence of hepatic, hematological, or renal dysfunction based on judgment of physician.
4. Subjects receiving treatment with topical steroids in areas to be stimulated.
5. Dermatopathology, skin hypersensitivity, or skin lesions in the area of measurements on the thigh and forearm.
6. Allergy to opioids.
7. Concomitant treatment with anticonvulsants, antidepressants, NMDA blockers, muscle relaxants, sedatives, other psychotropic drugs or opioids.
8. Is currently taking or has taken a monamine oxidase inhibitor (MAOI) drug within two weeks prior to study medication sessions.
9. Use of NSAIDs or acetaminophen within 36 hours of drug treatment sessions and/or use of caffeine or alcohol beginning 24 hours prior to the first drug treatment sessions.
10. Use of long-acting NSAIDs such as piroxicam or naproxen (Naprosyn) within 1 week of oral drug treatment sessions.
11. Heat pain detection thresholds above 47°C/116.6°F on the arm (see below).
12. Subjects who are not within following parameters for weight: between 110 and 200 pounds and between 20 and 30 using the Body Mass Index.
13. Subjects who are unable to read or speak English.
14. Diagnosis of insulin-requiring diabetes mellitus.
15. Current diagnosis of drug or alcohol abuse or history of opioid drug abuse
16. Use of opioids or alcohol while in study, confirmed by urine drug-screen at Session 1 and Session 2 and breathalyzer for alcohol at Sessions 2-6.
17. Neurological dysfunction or psychiatric disorder severe enough to interfere with assessment of pain and sensory systems.
18. Has received an investigational drug within 30 days prior to Study Visit 2 or is scheduled to receive another opioid medication during the course of this study.
19. Chronic pain condition requiring regular physician visits and prescription medication use on a daily basis.
20. Subjects who in the opinion of the investigator are considered unable to adhere to scheduled appointments, unlikely to comply with the study protocol, or who are unsuitable for any other reason.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2005-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To investigate the time course of development of analgesic tolerance (loss of pain relieving effect) to morphine on experimentally produced skin tenderness in healthy volunteers.

SECONDARY OUTCOMES:
To expand the knowledge about the analgesic (pain relieving) effects of opioids on experimentally induced pain and further validate the Brief Thermal Sensitization model as a tool for testing analgesic drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Petersen, MD, Principal Investigator — University of California, San Francisco; Michael C Rowbotham, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States